CLINICAL TRIAL: NCT02247947
Title: Proteomics to Identify Prognostic Markers After CPR and to Estimate Neurological Outcome
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Jochen Hinkelbein, Priv.-Doz. Dr. med., Universitätsklinikum Köln
Other Study IDs: 14-053
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Cardiac Arrest
Keywords: CPR
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- dead: Patients dead until day 20 (primary outcome measure)
- survivors: patients alive after day 20 (primary outcome measure)

SUMMARY:
Proteomics is used to identify prognostic markers after CPR. Additionally neurological outcome should be estimated by specific protein alterations and affections of pathways.

DETAILED DESCRIPTION:
Proteomics is used to identify prognostic markers after CPR, i.e. altered proteins on a 2G-gel. Additionally neurological outcome should be estimated by specific protein alterations and affections of pathways.

ELIGIBILITY:
Inclusion Criteria:

* cardiac arrest

Exclusion Criteria:

* trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cardiac arrest of non-trauma origin
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
death at day 20 | day 20

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hinkelbein, MD, Study Chair — UK Köln
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany